CLINICAL TRIAL: NCT03726229
Title: Development of a Reliable Means for Functional Assessment of Liver Performance After the Fontan Operation: Dual Cholate Clearance Assay
Brief Title: Cholate Clearance in Fontans
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: 829578
Record Dates: First submitted 2018-10-29; First posted 2018-10-31 (Actual); Last update posted 2022-06-10 (Actual); Status verified 2022-06

CONDITIONS: Fontan Procedure
Keywords: liver disease
MeSH Terms: conditions — Liver Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

GROUPS / COHORTS (1):
- Fontan patient: Cholate assay will be administered once to Fontan patients and blood specimens will be collected to analyze cholate clearance.
  Interventions: Device: Cholate assay

INTERVENTIONS:
Device: Cholate assay — Labeled oral and IV cholate will be administered once to the Fontan cohort and blood specimens will be collected at baseline and timepoints thereafter.
  Other Names: HepQuant assay

SUMMARY:
HepQuant is an assay to measure liver function in other forms of liver disease such as hepatitis C. It measures the ability of the liver to process an naturally occurring substance called cholate and has been shown to predict clinical outcomes in some patient populations.

The Fontan survivor is a patient who has undergone surgery or a series of surgeries that result in a functional single ventricle. The liver is particularly vulnerable to disease including congestion, fibrosis, and even cirrhosis. Currently liver function in the Fontan is not well-characterized and the HepQuant assay could help answer this question.

DETAILED DESCRIPTION:
A novel test called HepQuant® is an assay that has been used to measure liver function in other types of liver disease. In these populations, it is hoped that the assay may show more subtle or sub-clinical liver abnormalities that blood tests alone cannot detect. HepQuant® is a test that examines the ability of the liver to process a substance called cholate, which is a naturally occurring substance in the body. Cholate gets to the liver 2 ways: through the gut (by mouth) or through the blood (IV or intravenous). The test involves administering oral and IV cholate which is labeled. This label is NOT radioactive, but can act as an indicator/marker for evaluation purposes.

The purpose of this study is to develop a reliable means of measuring liver function in the Fontan survivor by examining cholate clearance. The investigators aim to 1) explore any association between level of cholate clearance and measurement of heart and liver function and 2) determine whether cholate clearance can predict clinical outcomes such as heart failure, ascites (development of fluid in the abdomen which can result from heart failure or liver failure), and need for heart transplant.

ELIGIBILITY:
Inclusion Criteria:

* s/p Fontan operation
* cardiac catheterization or cardiac MRI within 1 year of enrollment

Exclusion Criteria:

* pregnant or breastfeeding
* unable to comprehend and/or give informed consent
* sensitivity to human serum albumin, or its preparations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult Fontan survivors at least 18 years of age
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2022-05-25 (Actual); Study Completion 2022-05-25 (Actual)

PRIMARY OUTCOMES:
Hepatic cholate clearance | Through study completion, an average of 1 year
  D4-cholate and 13C-cholate clearance

SECONDARY OUTCOMES:
Incidence of adverse clinical outcomes | 5 years after cholate assay
  combined outcome of occurrence of any of the following: heart failure admission, clinically significant ascites, protein losing enteropathy, referral for cardiac transplantation, death

CONTACTS AND LOCATIONS:
Overall Officials: Yuli Kim, MD, Principal Investigator — University of Pennsylvania; Maarouf Hoteit, MD, Principal Investigator — Hospital of the University of Pennslyvania
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers

REFERENCES:
- [Derived] Kim YY, Nyman A, Huang YS, Tomlinson AZ, McRae MP, Everson GT, Vaikunth S, Rosenthal B, Rychik J, Hoteit MA. Alterations in Liver Perfusion in Adults With Fontan Circulation as Assessed by Dual Cholate Clearance. J Am Heart Assoc. 2025 Apr;14(7):e039479. doi: 10.1161/JAHA.124.039479. Epub 2025 Mar 21. PMID 40118791